CLINICAL TRIAL: NCT07246759
Title: NEUTROFLOW: Development and Validation of a Pan-cancer Neutrophil Biomarker Test for Predicting Clinical Benefit From Immunotherapy Based on Flow Cytometry Analysis of Blood Samples
Brief Title: Neutrophil Biomarker Test for Predicting Clinical Benefit From Immunotherapy Based on Flow Cytometry Analysis
Acronym: NEUTROFLOW
Status: Not yet recruiting | Type: Observational
Sponsor: OncoHost Ltd. (Industry)
Collaborators: European Institute of Oncology (Other); University Hospital Heidelberg (Other); Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor
Other Study IDs: NEUTROFLOW
Record Dates: First submitted 2025-11-16; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer (NSCLC); Melanoma (Skin Cancer); Triple Negative Breast Cancer (TNBC); RCC, Renal Cell Cancer; HNSCC
Keywords: Immunotherapy; Biomarker; Neutrophils; Flow Cytometry; Immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Triple Negative Breast Neoplasms; Carcinoma, Renal Cell; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood withdrawal at baseline before treatment initiation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients with stage IV or stage III unresectable non-small cell lung cancer (NSCLC): Patients with stage IV or stage III unresectable non-small cell lung cancer (NSCLC) treated with immune checkpoint inhibitors as a first-line treatment
  Interventions: Other: Blood sample collection
- Patients with stage IV or stage IIIb-d malignant melanoma: Patients with stage IV or stage IIIb-d malignant melanoma treated with immune checkpoint inhibitors as a first-line treatment
  Interventions: Other: Blood sample collection
- Patients with stage IV head and neck squamous cell carcinoma (HNSCC): Patients with stage IV head and neck squamous cell carcinoma (HNSCC) treated with immune checkpoint inhibitors as a first-line treatment
  Interventions: Other: Blood sample collection
- Patients with stage IV renal cell carcinoma (RCC): Patients with stage IV renal cell carcinoma (RCC) treated with immune checkpoint inhibitors as a first-line treatment
  Interventions: Other: Blood sample collection
- Patients with stage IV triple-negative breast cancer (TNBC): Patients with stage IV triple-negative breast cancer (TNBC) treated with immune checkpoint inhibitors as a first-line treatment
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — Blood sample collection prior treatment initiation

SUMMARY:
The NeutroFlow study is a multi-center clinical trial designed to develop a computational model that converts flow cytometry results into a prediction of clinical benefit. The study analyzes Ly6Ehi neutrophils in biological samples from patients treated with immune checkpoint inhibitors to evaluate their likelihood of benefiting from treatment. Blood samples are collected prior to treatment and used to support the ongoing development of the algorithm.

DETAILED DESCRIPTION:
The recent introduction of cancer immunotherapy based on immune checkpoint inhibitors (ICIs) has revolutionised the treatment landscape for a broad range of cancer types. However, response to ICIs varies widely between patients, with the majority experiencing resistance to therapy. Moreover, the increasing use of these costly drugs coupled with management of ICI-related toxicities creates a substantial economic burden. Current biomarker tests for determining eligibility for ICIs have limited predictive performance, and many require invasive tumour biopsies. Thus, novel (and preferentially non-invasive) biomarkers for predicting ICI clinical benefit are desperately needed for better guiding clinical decisions. NeutroFlow directly addresses this unmet need. The neutroFlow study is based on a comprehensive academic research describing a flow cytometry assay for measuring a novel predictive biomarker in the blood - Ly6Ehi neutrophil - that accurately predicts therapeutic benefit from ICIs, outperforming the approved PD-L1 biomarker.

The objective of the NeutroFlow study is to develop a clinical decision-support tool that includes an antibody panel for detecting Ly6Ehi neutrophils using standard flow cytometry (FC) and a computational model that converts the FC readout into a prediction of clinical benefit.

Patients will provide a single blood sample before starting treatment, and clinical data will be collected from their medical records.

In the first phase of the trial, blood sample data and clinical information will be used to develop the antibody panel and train the prediction algorithm. In the second phase, the algorithm will be validated by comparing its theoretical predictions with the patients' actual objective response rates.

ELIGIBILITY:
Inclusion Criteria:

• Patients newly diagnosed with advanced-stage/metastatic NSCLC, melanoma, HNSCC, RCC, or TNBC, who are due to receive first-line treatment with a PD-(L)1 inhibitor, either as monotherapy or in combination with other agents, according to current standard-of-care regimens, including (but not limited to) the following approved options: NSCLC. Monotherapy: Pembrolizumab, Atezolizumab, Cemiplimab. Combination: Pembrolizumab + chemotherapy; Nivolumab + Ipilimumab; Cemiplimab + chemotherapy; Atezolizumab + chemotherapy + Bevacizumab.

Melanoma. Monotherapy: Nivolumab, Pembrolizumab. Combination: Nivolumab + Ipilimumab; Nivolumab + Relatlimab.

HNSCC. Monotherapy: Pembrolizumab, Cemiplimab. Combination: Pembrolizumab + chemotherapy.

RCC. Combination only: Nivolumab + Ipilimumab; Nivolumab + Cabozantinib; Pembrolizumab + Lenvatinib or Axitinib; Avelumab + Axitinib.

TNBC. Combination only: Pembrolizumab + chemotherapy.

* Male or female aged at least 18 years
* ECOG PS: 0/1-2
* Normal hematologic, renal and liver function:

Absolute neutrophil count > 1500/mm³ Platelets > 100,000/mm³ Hemoglobin > 9 g/dL Creatinine concentration ≤ 1.4 mg/dL, or creatinine clearance > 40 mL/min, Total bilirubin < 1.5 mg/dL ALT + AST levels ≤ 3 times above the upper normal limit

Exclusion Criteria:

* Any concurrent and/or other active malignancy that has required systemic treatment within 2 years of the first dose of treatment.
* For NSCLC: presence of activating EGFR, ALK, ROS1, RET, NTRK alterations linked to an approved first-line targeted drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 600 treatment-naïve patients due to be treated with a first line regimen that includes PD- 1/PD-L1 inhibitors with the following diagnoses are planned to be enrolled in the study over a period of 3 years or as needed: 1. Stage IV or Stage III-unresectable NSCLC 2. Stage IV or Stage IIIb-d malignant melanoma 3. Stage IV HNSCC 4. Stage IV RCC 5. Stage IV TNBC
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Quantification of Ly6E high (Ly6Ehi) neutrophils in blood using the NeutroFlow flow cytometry assay | Baseline (up to 1 month before treatment initiation)
  Peripheral blood samples will be collected from patients up to 1 month prior to treatment initiation. Ly6Ehi neutrophil populations will be quantified using the NeutroFlow multiparametric flow cytometry assay
Prediction of clinical benefit rate using baseline Ly6Ehi neutrophils levels | Baseline (blood draw) to 6, 12, 18, and 24 months post treatment initiation
  The patients clinical benefit (CB) will be defined according to RECIST 1.1 criteria to one of the following categories: complete response (CR), partial response (PR), or stable disease (SD). Baseline Ly6Ehi neutrophil levels will be used as input in a computational predictive model to estimate the likelihood of CB for each patient. The model will be trained and validated with independent patient cohorts, using cross-validation and ROC AUC metrics to assess predictive performance. Sensitivity, specificity, positive predictive value, and negative predictive value will also be calculated. Predictions will be assessed at multiple timepoints: 6, 12, 18, and 24 months post-initiation of anti-PD-(L)1 therapy. Subgroup analyses will include age, sex, cancer type, disease stage, and treatment line.

SECONDARY OUTCOMES:
Clinical benefit rate across individual cancer types | Baseline to 6, 12, 18, and 24 months post treatment initiation (per indication)
  The clinical benefit rate described in Outcome 2 will be evaluated separately for each cancer indication (e.g., NSCLC, melanoma, HNSCC, RCC, TNBC) at several time points (6, 12, 18 and 24 months post treatment initiation). At least 50 patients per indication will be included to ensure adequate statistical power. ROC AUC values and predictive model performance will be computed for each subgroup. Additional exploratory analyses will examine potential modifiers, including tumor burden, prior therapies, and immune-related biomarkers, to evaluate heterogeneity of response
Clinical benefit rate by PD-(L)1 treatment regimen | Baseline to 6, 12, 18, and 24 months post treatment initiation
  The clinical benefit rate will be assessed across various anti-PD-(L)1 regimens, including monotherapy and combination protocols. Treatments are classified according to indication and line of therapy:
  NSCLC: Monotherapy: Pembrolizumab, Atezolizumab, Cemiplimab. Combination: Pembrolizumab + chemotherapy; Nivolumab + Ipilimumab; Cemiplimab + chemotherapy; Atezolizumab + chemotherapy + Bevacizumab.
  Melanoma: Monotherapy: Nivolumab, Pembrolizumab. Combination: Nivolumab + Ipilimumab; Nivolumab + Relatlimab.
  HNSCC: Monotherapy: Pembrolizumab, Cemiplimab. Combination: Pembrolizumab + chemotherapy.
  RCC: Combination only: Nivolumab + Ipilimumab; Nivolumab + Cabozantinib; Pembrolizumab + Lenvatinib or Axitinib; Avelumab + Axitinib.
  TNBC: Combination only: Pembrolizumab + chemotherapy.
  In cases where treatment changes occur during follow-up, two scenarios will be considered:
  1. the patient exits the analysis at the time of treatment change; or
  2. the new treatment marks a new baseline.
Correlation between Ly6Ehi neutrophil levels and PD-L1 status (TPS/CPS) | Baseline (PD-L1 and neutrophils assessed prior to treatment)
  Evaluation of the association between baseline Ly6Ehi neutrophil levels and PD-L1 expression in tumor tissue, measured as Tumor Proportion Score (TPS) and/or Combined Positive Score (CPS), depending on standard of care and assay availability. PD-L1 will be assessed by IHC using validated assays per standard of care. Subgroup analyses will explore correlations within different cancer types and treatment regimens. These analyses will provide insight into whether Ly6Ehi neutrophils complement or enhance PD-L1-based patient stratification.
Correlation between Ly6Ehi neutrophil levels and other clinical response-associated parameters | Baseline (clinical parameters collected prior to treatment)
  Exploratory analyses will assess correlations between baseline Ly6Ehi neutrophil levels and other parameters associated with immune checkpoint inhibitor (ICI) response, including Tumor Mutational Burden (TMB), Microsatellite Instability (MSI), Lactate Dehydrogenase (LDH), C-reactive protein (CRP), and ECOG performance status. Multivariate models and correlation analyses will evaluate whether Ly6Ehi neutrophils provide independent predictive value. Subgroup analyses will include cancer type, treatment regimen, and prior therapy exposure. This outcome will help determine the broader immunological and clinical context of Ly6Ehi neutrophil levels

CONTACTS AND LOCATIONS:
Locations (3):
- Heidelberg University Hospital, Heidelberg, Germany
- Intituto Europeo di Oncologia SRL, Milan, Italy
- Virgen Macarena University Hospital - Servicio Andaluz de Salud, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The clinical information and results generated as part of the study may be shared with other researchers and doctors, national and international regulatory agencies as well as in scientific repositories, always ensuring the necessary conditions of quality, security and confidentiality.

REFERENCES:
- [Background] Alturki NA. Review of the Immune Checkpoint Inhibitors in the Context of Cancer Treatment. J Clin Med. 2023 Jun 27;12(13):4301. doi: 10.3390/jcm12134301. PMID 37445336
- [Background] Man J, Millican J, Mulvey A, Gebski V, Hui R. Response Rate and Survival at Key Timepoints With PD-1 Blockade vs Chemotherapy in PD-L1 Subgroups: Meta-Analysis of Metastatic NSCLC Trials. JNCI Cancer Spectr. 2021 Jan 27;5(3):pkab012. doi: 10.1093/jncics/pkab012. eCollection 2021 Jun. PMID 34084999
- [Background] Martins F, Sofiya L, Sykiotis GP, Lamine F, Maillard M, Fraga M, Shabafrouz K, Ribi C, Cairoli A, Guex-Crosier Y, Kuntzer T, Michielin O, Peters S, Coukos G, Spertini F, Thompson JA, Obeid M. Adverse effects of immune-checkpoint inhibitors: epidemiology, management and surveillance. Nat Rev Clin Oncol. 2019 Sep;16(9):563-580. doi: 10.1038/s41571-019-0218-0. PMID 31092901
- [Background] Hurwitz JT, Vaffis S, Grizzle AJ, Nielsen S, Dodson A, Parry S. Cost-Effectiveness of PD-L1 Testing in Non-Small Cell Lung Cancer (NSCLC) Using In Vitro Diagnostic (IVD) Versus Laboratory-Developed Test (LDT). Oncol Ther. 2022 Dec;10(2):391-409. doi: 10.1007/s40487-022-00197-1. Epub 2022 May 13. PMID 35556235
- [Background] Lei Y, Li X, Huang Q, Zheng X, Liu M. Progress and Challenges of Predictive Biomarkers for Immune Checkpoint Blockade. Front Oncol. 2021 Mar 11;11:617335. doi: 10.3389/fonc.2021.617335. eCollection 2021. PMID 33777757
- [Background] Arora S, Velichinskii R, Lesh RW, Ali U, Kubiak M, Bansal P, Borghaei H, Edelman MJ, Boumber Y. Existing and Emerging Biomarkers for Immune Checkpoint Immunotherapy in Solid Tumors. Adv Ther. 2019 Oct;36(10):2638-2678. doi: 10.1007/s12325-019-01051-z. Epub 2019 Aug 13. PMID 31410780
- [Background] McKean WB, Moser JC, Rimm D, Hu-Lieskovan S. Biomarkers in Precision Cancer Immunotherapy: Promise and Challenges. Am Soc Clin Oncol Educ Book. 2020 May;40:e275-e291. doi: 10.1200/EDBK_280571. PMID 32453632
- [Background] Benguigui M, Cooper TJ, Kalkar P, Schif-Zuck S, Halaban R, Bacchiocchi A, Kamer I, Deo A, Manobla B, Menachem R, Haj-Shomaly J, Vorontsova A, Raviv Z, Buxbaum C, Christopoulos P, Bar J, Lotem M, Sznol M, Ariel A, Shen-Orr SS, Shaked Y. Interferon-stimulated neutrophils as a predictor of immunotherapy response. Cancer Cell. 2024 Feb 12;42(2):253-265.e12. doi: 10.1016/j.ccell.2023.12.005. Epub 2024 Jan 4. PMID 38181798

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT07246759/Prot_SAP_000.pdf